CLINICAL TRIAL: NCT02174744
Title: Concordance of Pain Detection in Patients by Doloplus® and Algoplus® Behavioural Scales.
Acronym: CALDOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr. Gisèle PICKERING (MCU, PH) Center of clinical pharmacology/CIC Inserm-1405 - Main investigator - Coordinating center (Unknown); Ms Joëlle DEVOT - Collaborator (Unknown); Dr Patrice RAT - Investigator (Unknown); Dr Chandra COLOM - Investigator (Unknown); Mr Dieudonné ENDOUGOU - Collaborator (Unknown); Dr Cyril GUILLAUME - Investigator (Unknown); Ms Nathalie ROUX - Collaborator (Unknown); Dr Yves PASSADORI - Investigator (Unknown); Ms Nathalie DANNENBERGER - Collaborator (Unknown); Dr Micheline MICHEL - Investigator (Unknown); Dr Sylvie CHAPIRO- Investigator (Unknown); Dr Jean-François VILLARD - Investigator (Unknown); Dr Bernard WARY- Investigator (Unknown); Dr Anne-Cécile BOURJAL - Investigator (Unknown); Dr Catherine BLUNTZ - Investigator (Unknown); Dr Françoise CAPRIZ - Investigator (Unknown); Dr Marie FLOCCIA - Investigator (Unknown); Dr Jérôme BOHATIER - Investigator (Unknown); Ms Linh NGUYEN PHUONG - Collaborator (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-0190
Record Dates: First submitted 2014-05-23; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Pain in Elderly Patients Having Communication Disorders.
Keywords: Pain in elderly patients having communication disorders; Numerical scale; Algoplus® scale; Doloplus® scale

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- numerical scale
  Interventions: Other: numeric pain rating scale

INTERVENTIONS:
Other: numeric pain rating scale

SUMMARY:
The pain of the elderly is often trivialized and ignored in spite of its high frequency: the chronic pain affects 50 % of the elderly living at home, 49 to 83 % of those living in institution and 80 % of this population at the end of life.

The evaluation of pain appeals to the same strategy as to the younger subject but with some specificities, related more to the pathologies associated with the ageing than to the real age. For that purpose, the investigators have self-assessment scales as the Numeric Pain Rating Scale which is adapted to estimate acute and chronic pains, but this scale presents a bias because, some patients do not express spontaneously their pain.

So behavioural scales were elaborated to solve the difficulties of detection and to care the pain of the elderly. The Algoplus® scale (5 items which takes less than one minute to be completed) whose objective is the observation of behavioural changes caused by the acute pain in elderly having communication disorders. The Doloplus® scale (30 items which allow in few minutes a good evaluation of pain) whose objective is the observation of behavioural changes caused by the chronic pain in elderly having communication impairments.

In practice, because of its popularity, the Algoplus® scale is widely used out of the specificity in which it has been validated. Practitioners, worried about this misuse, suggested to Doloplus® group, to test the concordance between the two behavioural scales in order to develop recommendations more targeted. The risk is that the use of the Algoplus® scale may underestimate pain that would have been detected by Doloplus® scale, and lead to under-treatment or non-treatment of pain in elderly having communication disorders.

This study aims to establish the concordance between these two scales to generate advices and recommendations to assess efficiently the pain in this vulnerable population.

The main objective of this study is to assess whether the use of Algoplus® scale is in good concordance with Doloplus® scale.

The secondary objective of this study is to assess the concordance with different levels of Algoplus® pain scale: (0-1), (2-3), (4-5).

DETAILED DESCRIPTION:
The physician investigator will identify and include patients in the study according to the inclusion criteria. Management of patients do not differ from the usual care in the service concerned. During the usual patient care, several pain assessments will be performed: Numeric Pain Rating Scale, MMSE score if the patient is able to communicate, Algoplus® scale and Doloplus® scale will be performed by doctors and/or caregivers without patient's participation. The patient will be assessed by two doctors and or caregivers (the time interval between the two assessments must be as short as possible).

In a first step, 48 hours after patient admission in the care service, a first doctor/caregiver will assess pain with Numeric Pain Rating Scale and evaluate MMSE score if it is possible and then assess pain with the Algoplus® scale. The results of the Numeric Pain Rating Scale, the Algoplus® scale and the MMSE score will be recorded in the medical record and in the study Case Report Form.

In a second step, less than 3 hours after the first assessment, a second doctor/caregiver will assess pain with the Doloplus® scale and the result will be recorded in the medical record and in the study Case Report Form.

The Case Report Form (containing demographic data, the history of pain, analgesics treatment, scores of Numeric Pain Rating Scale, MMSE, Algoplus® scale and Doloplus® scale) will be faxed to the Coordinating Center at Clermont-Ferrand in the day.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 65 or more years old
* Patients having communication disorders
* Hospitalization for at least 48 hours

Exclusion Criteria:

* Patients of less than 65 years

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Pain scores on Algoplus® and Doloplus® pain scales | at 48 hours after patients' admission in the care service.

SECONDARY OUTCOMES:
Different levels of Algoplus® pain scale: (0-1), (2-3), (4-5) | at 48 hours after patients' admission in the care service.

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France